CLINICAL TRIAL: NCT01512953
Title: Randomized Comparison of PPI Versus no PPI on Top of Standard Dose Clopidogrel Therapy in Patients Stratified Based on CYC2C19 Activity Via a Genetic Point of Care System.
Brief Title: Effect of Proton Pump Inhibitor on Residual Platelet Reactivity After Clopidogrel in Homogenous Genetic Strata
Acronym: GENIOUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Marco Valgimigli, MD, PhD, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEN-2011-1
Record Dates: First submitted 2012-01-15; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Stenting
Keywords: PPI; clopidogrel; 2C19; Lansoprazole
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- no PPI (No Intervention): Patients, stratified according to the genetic stratum, will be randomized not to take any PPI on top of clopidogrel
- PPI (Experimental): Patients stratified to the genetic stratum will be randomized to take PPI on top of clopidogrel
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole 30 mg once a day
  Arms: PPI

SUMMARY:
This study aims to prospectively assess whether there is an interaction between genetic status in terms of 2C19 activity and residual platelet reactivity after clopidogrel intake in patients who underwent coronary stenting for elective, urgent or emergent intervention.

DETAILED DESCRIPTION:
In managing patients who undergo percutaneous coronary intervention (PCI), rapid and predictable platelet inhibition for all patients is an important therapeutic goal. Determining the optimal dose of antiplatelet therapy to achieve this goal has been hampered by considerable interpatient variability in response to clopidogrel, which largely reflects gene polymorphism. Most of the evidence is centred around cytochrome 450 2C19.

A substudy of TRITON TIMI 38 has recently shown that among persons treated with clopidogrel, carriers of a reduced-function CYP2C19 allele had significantly lower levels of the active metabolite of clopidogrel, diminished platelet inhibition, and a higher rate of major adverse cardiovascular events, including stent thrombosis, than did noncarriers (N Engl J Med 2009;360:354-62). As a contrary, common functional CYP genetic variants do not affect active drug metabolite levels, inhibition of platelet aggregation, or clinical cardiovascular event rates in persons treated with prasugrel (Circulation. 2009 May 19;119(19):2553-60).

More recently, it has been shown that CYP2C19*17 carrier status is significantly associated with enhanced response to clopidogrel and an increased risk of bleeding. (Circulation. 2010;121:512-518). Whether CYP2C19*17 carrier status enhances response to prasugrel is unknown.

Attention has also been placed on a potential interaction observed between clopidogrel and the widely used proton pump inhibitors (PPIs).

The CYP2C19 isoform is the key enzyme in the metabolism of many of the PPIs, which are also inhibitors of the CYP2C19 isoenzyme in varying degrees. This is important because the antiplatelet effects of clopidogrel rely, to a degree, upon CYP2C19 activity. However, the recent COGENT study and sub-analysis of the TRITON-TIMI 38 have both apparently mitigated this concern. Nevertheless, it is unknown whether PPI can father blunt response to clopidogrel especially in patients carrying the loss of function 2C19 allele.

A recent review paper (Aliment Pharmacol Ther 31, 810-823) included 23 studies covering 93,278 patients. There was substantial heterogeneity in the meta-analyses of major cardiovascular events (19 studies, I2 = 79%) or myocardial infarction (12 studies, I2 = 77%). Analysis of propensity-matched or randomized trial participants showed no associated cardiovascular risk with PPIs, whereas other observational studies generally showed a significant association.

Thus, still today there is an emerging need for more studies, especially prospective randomized studies, to investigate the effect of individual PPI agents on clopidogrel's effectiveness. Such studies should also include a genetic component to stratify response based on the presence of reduced-function alleles of the CYP2C19 enzyme

ELIGIBILITY:
Inclusion Criteria: All comer patients undergoing PCI will be recruited on a consecutive basis.

• Patients will undergo screening before or soon after PCI depending on their clinical presentation as follows:

* STEMI patients will receive upstream treatment with 600 mg clopidogrel before PCI and will undergo screening for 2C19 status within 24 hours after treatment. Randomization will occur immediately thereafter.
* Stable and NSTEACS patients will be treated upstream with 600 mg clopidogrel and will undergo screening either before PCI or soon after (within 6 hours) revascularisation. In both scenarios randomization will occur immediately after the genotype status is known without any additional delay.

Exclusion Criteria:

1. Patients who can not give informed consent or have a life expectancy of < 1 year
2. Ongoing bleeding or bleeding diathesis or increase bleeding risk or history of bleeding in the last 2 months
3. Age > 90
4. Previous stroke or TIA or any intracranial pathology
5. Major surgery or trauma within the previous six weeks
6. Platelet count < 100.000 per cubic mm or HCT ,33% or Hb < 11 gm/dL
7. Subjects with an allergy or intolerance to prasugrel or to clopidogrel
8. Planned elective cardiac or non-cardiac surgery within 1 month.
9. Current or planned therapy with coumadin anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Maximal platelet aggregation at light transmission aggregometry after 20 μmol/l ADP | 30 days
  IPA expressed as maximal platelet aggregation (MPA) after 20 μmol/l ADP according to genetic stratum defined as follows: [(Poor metabolizers: 2C19*2+ and 2C19*17-); (intermediate metabolizers: wild type patients or its carrying both 2C19*2 and *170; (ultra metabolizers: 2c19*2- and 2C19*17+).
maximal platelet aggregation after 5 μmol/l ADP in PPI versus no PPI treated patients | 30 days
  Patients, stratified by genetic stratum, will be randomized to PPI or no PPI. We assume that that will be an interaction in the IPA after 5 μmol/l ADP at 30 days so that PPI will blunt responsiveness to clopidogrel in poor metabolizer patients only but in intermediate or ultra metabolizers.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ferrara, Ferrara, ER, Italy